CLINICAL TRIAL: NCT03529123
Title: A Randomized, 24-week, Controlled, Open Label, Parallel Arm, Multicenter Study Comparing the Efficacy and Safety of the Insulin Glargine/Lixisenatide Fixed Ratio Combination to Insulin Glargine in Type 2 Diabetes Patients, Inadequately Controlled on Basal Insulin With or Without Metformin
Brief Title: Efficacy and Safety of the Insulin Glargine/Lixisenatide Fixed Ratio Combination Versus Insulin Glargine in Patients With Type 2 Diabetes (LixiLan-India)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INSLIL08556; U1111-1200-1162 (Other: UTN)
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide; Metformin; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tested Drug (Experimental): Insulin glargine/lixisenatide fixed ratio combination (FRC)
  Interventions: Drug: INSULIN GLARGINE/LIXISENATIDE (HOE901/AVE0010); Drug: Metformin; Drug: Insulin Glulisine (HMR1964)
- Control Drug (Active Comparator): Insulin glargine (Lantus®)
  Interventions: Drug: INSULIN GLARGINE (HOE901); Drug: Metformin; Drug: Insulin Glulisine (HMR1964)

INTERVENTIONS:
Drug: INSULIN GLARGINE/LIXISENATIDE (HOE901/AVE0010) — Pharmaceutical form: Injection
  Route of administration: Subcutaneous
  Other Names: Soliqua, Insulin Glargine/Lixisenatide Fixed Ratio Combination
  Arms: Tested Drug
Drug: INSULIN GLARGINE (HOE901) — Pharmaceutical form: Injection
  Route of administration: Subcutaneous
  Other Names: Lantus®
  Arms: Control Drug
Drug: Metformin — Pharmaceutical form: Tablet
  Route of administration: Oral
Drug: Insulin Glulisine (HMR1964) — Pharmaceutical form: Injection
  Route of administration: Subcutaneous
  Other Names: Apidra

SUMMARY:
Primary Objective:

To demonstrate the superiority of the insulin glargine/lixisenatide fixed ratio combination (FRC) to insulin glargine by demonstrating change in glycosylated hemoglobin (HbA1c).

Secondary Objectives:

* To assess the effects of the FRC in comparison with insulin glargine on:
* Percentage of patients reaching HbA1c targets (<7% );
* Glycemic control in relation to a meal as evaluated by 2-hour Post-prandial Plasma Glucose; (PPG);
* Body weight
* Fasting Plasma Glucose (FPG);
* Percentage of patients reaching HbA1c targets of <7% with no body weight gain and no hypoglycemia (as defined in the evaluation criteria);
* 7-point Self-Monitoring Plasma Glucose (SMPG) profile;
* Insulin glargine dose.
* To assess the safety and tolerability in each treatment group.

DETAILED DESCRIPTION:
The maximum study duration per patient is 33 weeks.

ELIGIBILITY:
Inclusion criteria :

* Patients with type 2 diabetes mellitus (T2DM) diagnosed for at least 1 year before the screening visit,
* At screening:
* Age should be ≥ 18 years of age to < 65 years;
* Glycosylated hemoglobin (HbA1c) at screening visit ≥ 7.5% or ≤ 10%;
* Body mass index (BMI) ≥ 19 kg/m2 and ≤ 40 kg/m2.
* Patients who have been treated with a basal insulin for at least 6 months before the screening visit, and who have been on a stable basal insulin regimen (ie, type of insulin and time/frequency of the injection), for at least 3 months before the screening visit. The stable total daily dose should be within the range of 15-40 U, both inclusive, on the day of screening, but individual fluctuations of ± 20% within 2 months prior to screening are acceptable.

Exclusion criteria:

* Use of oral or injectable glucose-lowering agents other than those stated in the inclusion criteria in the 3 months before screening.
* Previous use of insulin regimen other than basal insulin eg, prandial or pre-mixed insulin (Note: Short term treatment due to intercurrent illness including gestational diabetes is allowed at the discretion of the investigator).
* For patients taking metformin, any contraindication to metformin use, according to local labeling.
* For patient not treated with metformin at screening: severe renal function impairment with an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2 or end-stage renal disease.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic condition that predisposes to MTC (eg, multiple endocrine neoplasia syndromes).
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including (but not limited to): gastroparesis, unstable (ie, worsening) or not controlled (ie, prolonged nausea and vomiting) gastroesophageal reflux disease requiring medical treatment, within 6 months prior to the time of screening visit; or history of surgery affecting gastric emptying.
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy has been performed), pancreatitis during previous treatment with incretin therapies, chronic pancreatitis, pancreatectomy.
* Average insulin glargine daily dose <20 U or >50 U calculated for the last 3 days before Visit 6.
* Amylase and/or lipase >3 upper limit normal (ULN) at Visit 5 (Week -1).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 247 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | From baseline to Week 24
  Mean change in glycosylated hemoglobin (HbA1c) from baseline to Week 24

SECONDARY OUTCOMES:
Patients with HbA1c <7% | At Week 24
  Number of patients reaching HbA1c <7 % at the end of Week 24
Change in 2-hour Post prandial glucose (PPG) | From baseline to Week 24
  Change in 2-hour PPG from baseline to Week 24
Change in body weight | From baseline to Week 24
  Change in body weight from baseline to Week 24
Patients with HbA1c <7% with no body weight gain and no hypoglycemia | At Week 24
  Number of patients reaching HbA1c <7% with no body weight gain and no hypoglycemia at the end of Week 24
Change in Fasting Plasma Glucose | From baseline to Week 24
  Mean change in FPG from baseline to Week 24
Adverse events (AE) | Up to 33 weeks
  Number of AEs
Patients with HbA1c <7% with no body weight gain | At Week 24
  Number of patients reaching HbA1c <7% with no body weight gain at the end of Week 24
Change in SMPG profiles | From baseline to Week 24
  Change in 7-point self-monitoring plasma glucose (SMPG) profiles from baseline to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- India (13):
  - Investigational Site Number 01, Bangalore
  - Investigational Site Number 012, Belagavi
  - Investigational Site Number 013, Chennai
  - Investigational Site Number 017, Coimbatore
  - Investigational Site Number 06, Hyderabad
  - Investigational Site Number 07, Hyderabad
  - Investigational Site Number 08, Jaipur
  - Investigational Site Number 04, Kolkata
  - Investigational Site Number 018, Lucknow
  - Investigational Site Number 014, Madurai
  - Investigational Site Number 05, Nashik
  - Investigational Site Number 010, New Delhi
  - Investigational Site Number 016, Pune

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org